CLINICAL TRIAL: NCT06318611
Title: Sleep Patterns and Chronotype Among Children and Adolescents With Type 1 Diabetes Compared to Case-control Peers Without Diabetes
Brief Title: Sleep Patterns and Chronotype in Children With and Without Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Koç University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2022.575
Record Dates: First submitted 2024-02-19; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Type1diabetes; Sleep; Chronotype
Keywords: type 1 diabetes; chronotype; continuous glucose monitoring; glycemic variability; sleep health; sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sleep; Chronotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Children and adolescents diagnosed with type 1 diabetes aged between 6 to 18 years
  Interventions: Other: sleep, chronotype
- Control group: Children and adolescents without type 1 diabetes between the ages of 6 and 18.
  Interventions: Other: sleep, chronotype

INTERVENTIONS:
Other: sleep, chronotype — Our objectives were to compare sleep health composite dimensions, and chronotype in children and adolescents with and without T1D, and to explore relationship between sleep and glycemic variability in T1D.

SUMMARY:
Type 1 diabetes (T1D) is one of the most common chronic childhood diseases. Recent studies have highlighted the strong association between type 1 diabetes and sleep health problems. Sleep problems have been reported to include sleep onset, sleep maintenance, frequent nighttime awakenings, and daytime sleepiness. Studies show that children with T1D sleep significantly less than their peers without diabetes, and that this is associated with poorer glycemic control in type 1 diabetes due to impaired glucose metabolism.

This study aimed to compare sleep health composite dimensions and chronotype in children and adolescents with and without T1D, and to explore the relationship between sleep and glycemic variability in T1D.

The study was designed as a prospective observational case-control study. The estimated sample size is calculated as 168.

The sleep health composite dimensions were measured using actigraphy, sleep diaries, and self- or parental reports. Sleep disturbance will be assessed using the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) Level 2-Sleep Disturbance Scale Short Form, and the Children's Chronotype Questionnaire will be used to determine the chronotype. Sleep/wake patterns were also assessed using sleep diaries. Glycemic variability was assessed using continuous glucose monitoring (CGM) device parameters.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is one of the most common chronic diseases in childhood. The prevalence of T1D in Turkey is reported to be 0.75%. Recent studies draw attention to the close relationship between type 1 diabetes and sleep problems. It has been suggested that sleep duration is insufficient and sleep quality is impaired in patients with T1D. Sleep problems have been reported to include sleep onset, sleep maintenance, frequent nighttime awakenings, and daytime sleepiness. Conditions such as nocturnal glycemic variability and fear of hypoglycemia specific to patients with T1D, alarms from devices such as continuous glucose monitors and pumps used in diabetes management, anxiety, stress and depressive symptoms associated with diabetes, and treatment that may sometimes last throughout the night are possible factors that adversely affect the sleep health of people with diabetes. Studies show that children with T1D sleep significantly less than their peers without diabetes and that this is associated with poorer glycemic control in type 1 diabetes due to impaired glucose metabolism. The American Diabetes Association (ADA) has emphasized that sleep health should be included in the routine assessment of people with diabetes by 2022.

This study aimed to compare sleep health composite dimensions and chronotype in children and adolescents with and without T1D, and to explore the relationship between sleep and glycemic variability in T1D.

The study was designed as a prospective observational case-control study. The estimated sample size is calculated as 168.

The sleep health composite dimensions were measured using actigraphy, sleep diaries, and self- or parental reports. This composite evaluates various dimensions of sleep, including regularity, satisfaction, alertness, timing, efficiency, and duration. Each dimension is assigned a code of '1' for 'good' and '0' for 'poor.' The sleep health composite is designed so that a higher score indicates better overall sleep health.

Sleep disturbances were assessed using the DSM-5 Level 2-Sleep Disturbance Scale Short Form. The DSM-5 Level 2-Sleep Disorders Scale short form was used to evaluate sleep disturbances. It is an 8-item scale that specifically evaluates sleep disorders in children and adolescents, within the past 7 days. Each item is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often, and 5=always). The total score ranges from 8 to 40 points, with higher scores indicating more severe sleep disturbances. Sleep/wake patterns were also assessed using sleep diaries.

The Childhood Chronotype Questionnaire was used to evaluate the chronotype in children. This 27-item questionnaire was developed for Turkish children in the light of the Munich Chronotype Questionnaire and the Mornings-Evenings Questionnaire. The chronotypes were classified as morning, intermediate and evening types, corresponding scores of ≤23, 24-32 and ≥33. The child form of the Childhood Chronotype Questionnaire was completed by the parent and the adolescent form was completed by the adolescent.

Glycemic variability was assessed using continuous glucose monitoring (CGM) device parameters. Glycemic variability was evaluated using the J index to assess the effectiveness of glycemic control (calculated as 0.001 × (mean + SD)), the low blood glucose index (LBGI) to evaluate the risk of hypoglycemia, the high blood glucose index (HBGI) to determine the likelihood of hyperglycemia, and the Coefficient of Variation (CV). The Coefficient of Variation expresses the percentage variation in blood glucose levels, with a CV ≤36% indicating a stable glucose profile and a CV >36% indicating an unstable glucose profile. For 24-hour continuous glucose monitoring, the targeted percentages of time were >70% at 70-180 mg/dl for glycemic control, <4% at <70 mg/dl for hypoglycemia, <1% at <54 mg/dl for severe hypoglycemia, <25% at >180 mg/dl for hyperglycemia and <5% at >250 mg/dl for severe hyperglycemia. The hemoglobin A1c level is also used for glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 to 18 years
* Use of continuous glucose monitor system

Exclusion Criteria:

* Acute medical condition that can impact sleep (diabetic ketoacidosis, cold, influenza)
* Diagnosed neurodevelopmental or behavioral conditions like autism spectrum disorder or Attention Deficit/Hyperactivity Disorder
* Diagnosed sleep disorder (Obstructive Sleep Apnea)
* Current use of medications that can impact sleep (diphenhydramine)

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents diagnosed with and without type 1 diabetes aged between 6 to 18 years
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Sleep health composite | Prospective, up to 24 weeks
  The sleep health composite dimensions were measured using actigraphy, sleep diaries, and self- or parental reports. This composite evaluates various dimensions of sleep, including regularity, satisfaction, alertness, timing, efficiency, and duration. Sleep disturbances were assessed using the DSM-5 Level 2-Sleep Disturbance Scale Short Form. The DSM-5 Level 2-Sleep Disorders Scale short form was used to evaluate sleep disturbances. It is an 8-item scale that specifically evaluates sleep disorders in children and adolescents within the past 7 days. Each item is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often, and 5=always). The total score ranges from 8 to 40 points, with higher scores indicating more severe sleep disturbances.
Chronotype | Prospective, up to 24 weeks
  Chronotype was evaluated by the Children's Chronotype Questionnaire. The Childhood Chronotype Questionnaire was used to evaluate the chronotype in children. This 27-item questionnaire was developed for Turkish children in the light of the Munich Chronotype Questionnaire and the Mornings-Evenings Questionnaire. The chronotypes were classified as morning, intermediate and evening types, corresponding scores of ≤23, 24-32 and ≥33. The child form of the Childhood Chronotype Questionnaire was completed by the parent and the adolescent form was completed by the adolescent.

SECONDARY OUTCOMES:
Glycemic variability | Prospective, up to 24 weeks
  Glycemic variability was assessed using continuous glucose monitoring device parameters. Glycemic variability was evaluated using the J index to assess the effectiveness of glycemic control, the low blood glucose index (LBGI) to evaluate the risk of hypoglycemia, the high blood glucose index (HBGI) to determine the likelihood of hyperglycemia, and the Coefficient of Variation.
Glycemic control | Prospective, up to 24 weeks
  For 24-hour continuous glucose monitoring, the targeted percentages of time were >70% at 70-180 mg/dl for glycemic control, <4% at <70 mg/dl for hypoglycemia, <1% at <54 mg/dl for severe hypoglycemia, <25% at >180 mg/dl for hyperglycemia and <5% at >250 mg/dl for severe hyperglycemia. The hemoglobin A1c level is also used for glycemic control.

CONTACTS AND LOCATIONS:
Locations (1):
- Necla İpar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ipar N, Boran P, Baris HE, Us MC, Aygun B, Haliloglu B, Baygul A, Mutlu GY, Bereket A, Hatun S. The sleep health composite and chronotype among children and adolescents with type 1 diabetes compared to case-control peers without diabetes. J Clin Sleep Med. 2025 May 1;21(5):825-834. doi: 10.5664/jcsm.11558. PMID 39789979